CLINICAL TRIAL: NCT00425360
Title: A Prospective, Phase III, Controlled, Multicentre, Randomised Clinical Trial Comparing Combination Gemcitabine and Capecitabine Therapy With Concurrent and Sequential Chemoimmunotherapy Using a Telomerase Vaccine in Locally Advanced and Metastatic Pancreatic Cancer [TELOVAC]
Brief Title: Gemcitabine and Capecitabine With or Without Vaccine Therapy in Treating Patients With Locally Advanced or Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Royal Liverpool University Hospital (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000528021; CRUK-TELOVAC-V4; EUDRACT-2006-000461-10; EU-20683; ISRTCN43482138
Record Dates: First submitted 2007-01-19; First posted 2007-01-23 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2009-05

CONDITIONS: Pancreatic Cancer
Keywords: stage III pancreatic cancer; stage IV pancreatic cancer; duct cell adenocarcinoma of the pancreas; recurrent pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — sargramostim; Capecitabine; Gemcitabine

INTERVENTIONS:
Biological: sargramostim
Biological: telomerase peptide vaccine GV1001
Drug: capecitabine
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Vaccines made from peptides may help the body build an effective immune response to kill tumor cells. Giving more than one drug (combination chemotherapy) together with vaccine therapy may kill more tumor cells. It is not yet known whether chemotherapy is more effective with or without vaccine therapy in treating pancreatic cancer.

PURPOSE: This randomized phase III trial is studying gemcitabine, capecitabine, and vaccine therapy to see how well they work compared with gemcitabine and capecitabine alone in treating patients with locally advanced or metastatic pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of telomerase peptide vaccine GV1001 when administered concurrently or sequentially with gemcitabine hydrochloride and capecitabine, in terms of survival, in patients with locally advanced or metastatic pancreatic cancer.

Secondary

* Determine the safety of this regimen in these patients.
* Assess the immunogenicity of this regimen in these patients.
* Determine the time to progression in patients treated with this regimen.
* Determine the quality of life of patients treated with this regimen.
* Determine the clinical benefit response in patients treated with this regimen.
* Determine the objective response rate in patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.
* Determine the survival and response by delayed-type hypersensitivity in patients treated with this regimen.

OUTLINE: This is a prospective, controlled, randomized, open-label, multicenter study. Patients are stratified according to stage of disease (locally advanced vs metastatic) and ECOG performance status (0 vs 1 vs 2). Patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15 and oral capecitabine twice daily on days 1-21. Treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive gemcitabine hydrochloride and capecitabine as in arm I. Treatment repeats every 4 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity. Patients then receive sargramostim (GM-CSF) intradermally (ID) and telomerase peptide vaccine GV1001 ID on days 1, 3, and 5 in week 9, once a week in weeks 10-12 and 14, and then once a month in the absence of disease progression or unacceptable toxicity. Patients who develop disease progression while on vaccine therapy, discontinue vaccine therapy and then restart treatment with gemcitabine hydrochloride and capecitabine. Patients receive gemcitabine hydrochloride and capecitabine as above and continue treatment in the absence of further disease progression or unacceptable toxicity.
* Arm III: Patients receive gemcitabine hydrochloride and capecitabine as in arm I. Patients also receive GM-CSF ID and telomerase peptide vaccine GV1001 ID on days 1, 3, and 5 in week 1, once weekly in weeks 2, 3, 4 and 6, and then once a month in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline and at 8 weeks and then every 12 weeks during study treatment.

After completion of study treatment, patients are followed every 3 months.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 1,110 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed pancreatic ductal adenocarcinoma or undifferentiated carcinoma of the pancreas

  * Locally advanced or metastatic disease precluding curative surgical resection
* Unidimensionally measurable disease by CT scan
* No intracerebral metastases or meningeal carcinomatosis

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy > 3 months
* WBC > 3,000/mm³
* Absolute neutrophil count > 1,500/mm³
* Platelet count > 100,000/mm³
* Bilirubin < 2.0 mg/dL
* Creatinine clearance > 50 mL/min
* No medical or psychiatric condition that would preclude giving informed consent
* No clinically significant serious disease or organ system disease not currently controlled on present therapy
* No uncontrolled angina pectoris
* Not pregnant or nursing
* Fertile patients must use a condom and ≥ 1 other form of contraception during and for 1 year after completion of study treatment
* No other malignancies or invasive cancers within the past 5 years except for adequately treated basal cell carcinoma of the skin or carcinoma in situ of the cervix
* No known malabsorption syndrome
* No known hypersensitivity to any of the investigational agents
* No dihydropyrimidine dehydrogenase deficiency

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy
* No radiotherapy within the past 4 weeks
* No concurrent medications that could affect immunocompetence (e.g., chronic treatment with long-term steroids or other immunosuppressants for unrelated condition)

  * Concurrent short-term steroids for palliation of cancer-related symptoms allowed
* No other concurrent investigational drugs or cytotoxic agents
* No other concurrent immunotherapy (e.g., immunosuppressants or chronic use of systemic corticosteroids) or chemotherapy for another tumor in patients receiving telomerase peptide vaccine GV1001

  * Concurrent low-dose corticosteroids may be allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1110 (Estimated)
Dates: Start 2006-09; Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Survival at 1 year

SECONDARY OUTCOMES:
Time to progression
Quality of life as assessed by the European Organization for Research and Treatment of Cancer (EORTC)-Quality of Life (QLQ) C30 questionnaire and the European Study group for Pancreatic Cancer-QLQ questionnaire
Clinical benefit response
Objective response rate as assessed by RECIST criteria
Toxicity as assessed by NCI CTCAE version 3
Survival and response as assessed by delayed-type hypersensitivity

CONTACTS AND LOCATIONS:
Overall Officials: Gary W. Middleton, Study Chair — St. Luke's Cancer Centre at Royal Surrey County Hospital
Locations (45):
- United Kingdom (45):
  - North Devon District Hospital, Barnstaple, England
  - Basingstoke and North Hampshire NHS Foundation Trust, Basingstoke, England
  - Pilgrim Hospital, Boston, England
  - Royal Bournemouth Hospital, Bournemouth, England
  - Sussex Cancer Centre at Royal Sussex County Hospital, Brighton, England
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Addenbrooke's Hospital, Cambridge, England
  - Darent Valley Hospital, Dartford Kent, England
  - Dorset County Hospital, Dorchester, England
  - Royal Devon and Exeter Hospital, Exeter, England
  - St. Luke's Cancer Centre at Royal Surrey County Hospital, Guildford, England
  - Huddersfield Royal Infirmary, Huddersfield, West Yorks, England
  - Ipswich Hospital, Ipswich, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Royal Liverpool University Hospital, Liverpool, England
  - Saint Bartholomew's Hospital, London, England
  - Cancer Research UK Clinical Groups at Guy's King's & St. Thomas' Hospitals, London, England
  - St. George's Hospital, London, England
  - Royal Marsden - London, London, England
  - Christie Hospital, Manchester, England
  - Clatterbridge Centre for Oncology, Merseyside, England
  - James Cook University Hospital, Middlesbrough, England
  - Northern Centre for Cancer Treatment at Newcastle General Hospital, Newcastle upon Tyne, England
  - James Paget Hospital, Norfolk, England
  - Mount Vernon Cancer Centre at Mount Vernon Hospital, Northwood, England
  - Norfolk and Norwich University Hospital, Norwich, England
  - Nottingham City Hospital, Nottingham, England
  - Churchill Hospital, Oxford, England
  - Peterborough Hospitals Trust, Peterborough, England
  - Dorset Cancer Centre, Poole Dorset, England
  - Portsmouth Oncology Centre at Saint Mary's Hospital, Portsmouth Hants, England
  - Conquest Hospital, Saint Leonards-on-Sea, England
  - Salisbury District Hospital, Salisbury, England
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - Wexham Park Hospital, Slough, Berkshire, England
  - Royal Marsden - Surrey, Sutton, England
  - Torbay Hospital, Torquay Devon, England
  - Royal Cornwall Hospital, Truro, Cornwall, England
  - Worthing Hospital, Worthing, England
  - Yeovil District Hospital, Yeovil, England
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Beatson West of Scotland Cancer Centre, Glasgow, Scotland
  - Glan Clwyd Hospital, Rhyl, Denbighshire, Wales
  - Wrexham Maelor Hospital, Wrexham, Wales